CLINICAL TRIAL: NCT00485927
Title: The Effects of Stress on the Clinical Performance of Residents in Simulated Trauma Scenarios
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Toronto (Other)
Collaborators: The Physicians' Services Incorporated Foundation (Other)
Allocation: Not Applicable | Model: Single Group | Masking: Double | Purpose: Health Services Research
Other Study IDs: 07-10
Record Dates: First submitted 2007-06-11; First posted 2007-06-13 (Estimated); Last update posted 2007-06-13 (Estimated); Status verified 2007-06

CONDITIONS: Trauma; Stress
Keywords: Trauma; Stress; Simulation
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: stress

SUMMARY:
Medical practice & training are inherently stressful situations. However, the effects of stress on educational & clinical performance are not well defined. The purpose of the current study is to examine the effects of stress on performance of residents in simulated trauma scenarios. The hypothesis is: 1) acutely stressful scenarios will be appraised as threat by residents and result in elevations of heart rate and salivary cortisol; 2) increased subjective & physiological stress will result in impairments in performance; and 3) greater stress responses will result in greater clinical impairments.

ELIGIBILITY:
Inclusion Criteria:

* University of Toronto General Surgery & Emergency medicine residents

Exclusion Criteria:

* No ATLS training
* Residents from other programs

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2007-04

PRIMARY OUTCOMES:
performance - global ratings
performance - ANTS
performance - checklists

CONTACTS AND LOCATIONS:
Overall Officials: Adrian M Harvey, MD, Principal Investigator — University of Toronto, University Health Network; Avery B Nathans, MD, PhD, Study Chair — University of Toronto, St. Michael's Hospital; Vicki Leblanc, PhD, Study Director — University of Toronto
Locations (1):
- St Michaels' Hospital, Toronto, Ontario, Canada